CLINICAL TRIAL: NCT02261220
Title: A Phase I Study of MEDI4736 (Anti-PD-L1 Antibody) in Combination With Tremelimumab (Anti-CTLA-4 Antibody) in Subjects With Advanced Solid Tumors
Brief Title: A Phase 1 Study of MEDI4736 in Combination With Tremelimumab in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4190C00010
Record Dates: First submitted 2014-10-02; First posted 2014-10-10 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Advanced Solid Tumors
Keywords: advanced solid tumors; durvalumab; tremelimumab
MeSH Terms: interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MEDI4736 + Tremelimumab (Experimental): Subjects with multiple tumor types.
  Interventions: Biological: MEDI4736; Biological: tremelimumab

INTERVENTIONS:
Biological: MEDI4736 — MEDI4736 is administered by IV infusion in combination with tremelimumab
Biological: tremelimumab — Tremelimumab is administered by IV infusion in combination with MEDI4736

SUMMARY:
This is a multicenter, open-label, dose-exploration and dose-expansion study to evaluate the safety, tolerability, antitumor activity, PK and immunogenicity of MEDI4736 in combination with tremelimumab in subjects with select advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* 18 years and older
* Histologic confirmation of advanced solid tumors
* Subjects must have recurrent/metastatic disease and may have been previously treated in the recurrent/metastatic setting.

Exclusion Criteria:

* Any concurrent chemotherapy, immune-mediated therapy or biologic or hormonal therapy for cancer treatment
* Active or prior documented autoimmune disease within the past 2 years
* Current or prior use of immunosuppressive medication within 14 days with some exceptions.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting adverse events | Screening through 15 months after the last subject enters re-treatment
Number of subjects reporting serious adverse events | Screening through 15 months after the last subject enters re-treatment
Number of subjects experiencing a dose-limiting toxicity | First dose of study medication through 4 weeks after the first dose of study medication
Change from Baseline in laboratory evaluations | Screening through 3 months after the last dose of study medication
Change from Baseline in vital signs | Screening through 3 months after the last dose of study medication
Change from Baseline in electrocardiogram evaluations | Screening through 3 months after the last dose of study medication
Overall Response Rate in Select Tumor Types | First dose of study medication through 15 months after the last subject enters re-treatment

SECONDARY OUTCOMES:
Overall Response Rate | First dose of study medication through 15 months after the last subject enters re-treatment
Disease Control Rate | First dose of study medication through 15 months after the last subject enters re-treatment
Duration of Response | First dose of study medication through 15 months after the last subject enters re-treatment
Progression-Free Survival | First dose of study medication through 15 months after the last subject enters re-treatment
Overall Survival | First dose of study medication through 15 months after the last subject enters re-treatment
Individual MEDI4736 concentrations | First dose of MEDI4736 through 3 months after the last dose of study medication
Individual tremelimumab concentrations | First dose of tremelimumab through 3 months after the last dose of study medication
MEDI4736 area under the concentration-curve | First dose of MEDI4736 through 3 months after the last dose of study medication
Tremelimumab area under the concentration-curve | First dose of tremelimumab through 3 months after the last dose of study medication
Number of subjects that develop detectable antidrug antibodies to MEDI4736 | First dose of MEDI4736 through 3 months after the last dose of study medication
Number of subjects that develop antidrug antibodies to tremelimumab | First dose of tremelimumab through 3 months after the last dose of study medication

OTHER OUTCOMES:
Change in Biomarkers | Screening through 3 months following the last dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (62):
- United States (26):
  - Research Site, Scottsdale, Arizona
  - Research Site, Duarte, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Whittier, California
  - Research Site, Aurora, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Miami Beach, Florida
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, Ann Arbor, Michigan
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Seattle, Washington
- Canada (4):
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- France (9):
  - Research Site, Angers
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Pierre-Bénite
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Villejuif
- Germany (3):
  - Research Site, Jena
  - Research Site, Münster
  - Research Site, Tübingen
- Israel (4):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Tel Aviv
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Tilburg
- South Korea (5):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Gwangju
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Valencia
- United Kingdom (5):
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Middlesbrough
  - Research Site, Oxford

REFERENCES:
- [Derived] Zhang Q, Luo J, Wu S, Si H, Gao C, Xu W, Abdullah SE, Higgs BW, Dennis PA, van der Heijden MS, Segal NH, Chaft JE, Hembrough T, Barrett JC, Hellmann MD. Prognostic and Predictive Impact of Circulating Tumor DNA in Patients with Advanced Cancers Treated with Immune Checkpoint Blockade. Cancer Discov. 2020 Dec;10(12):1842-1853. doi: 10.1158/2159-8290.CD-20-0047. Epub 2020 Aug 14. PMID 32816849